CLINICAL TRIAL: NCT00981253
Title: Enhancing Standard Cardiac Rehabilitation With Stress Management Training in Patients With Heart Disease
Brief Title: Stress Management and Biomarkers of Risk in Cardiac Rehabilitation
Acronym: ENHANCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015896; R01HL093374-01A2 (NIH)
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Coronary Heart Disease
Keywords: Stress Management Training; Cardiac Rehabilitation; Stress; Depression
MeSH Terms: conditions — Coronary Disease; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMT-enhanced Cardiac Rehabilitation (Experimental): Standard exercise-based cardiac rehabilitation with weekly stress management training for 12 weeks.
  Interventions: Behavioral: SMT-enhanced Cardiac Rehabilitation
- Standard Cardiac Rehabilitation (Active Comparator): Standard cardiac rehabilitation consisting of supervised exercise for 12 weeks.
  Interventions: Behavioral: Standard Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: SMT-enhanced Cardiac Rehabilitation — Standard exercise-based cardiac rehabilitation, three times per week, enhanced with weekly stress management training for 12 weeks.
  Arms: SMT-enhanced Cardiac Rehabilitation
Behavioral: Standard Cardiac Rehabilitation — Supervised exercise, three times per week, for 12 weeks.
  Arms: Standard Cardiac Rehabilitation

SUMMARY:
The purpose of this study is to assess the extent to which combining exercise and stress management training (SMT) is more effective at improving biomarkers in vulnerable cardiac patients compared to exercise-based cardiac rehabilitation alone.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the leading cause of death in the United States and in roughly half the cases its first clinical manifestations, myocardial infarction (MI) or sudden cardiac death (SCD), are fatal. There is considerable evidence that "stress" plays a significant and independent role in the occurrence of CHD and its complications. This evidence has provided the rationale for developing interventional strategies to reduce stress in susceptible individuals in order to modify the natural history of these clinical events. There are now promising data to suggest that stress management training (SMT) is one such approach, and that SMT can have beneficial effects on psychosocial and medical outcomes. However, many of the randomized clinical trials (RCTs) employing stress management approaches in CHD patients have had important methodological limitations and several of the larger RCTs have failed to demonstrate a benefit for SMT over usual care, raising questions about the value of SMT for patients with CHD. Reliance on "hard" clinical endpoints is problematic because studies require such large sample sizes that they are logistically difficult to conduct and are prohibitively expensive. The use of intermediate pathophysiologic endpoints that have been shown independently to be associated with increased risk represents a novel and exciting opportunity to examine the added value of SMT in exercise-based cardiac rehabilitation (CR) compared to CR without SMT on key biomarkers of risk in vulnerable CHD patients.

This 12-week study will enroll adults with stable CHD who are eligible for CR. Participants will be randomly assigned to either standard cardiac rehabilitation or standard cardiac rehabilitation enhanced with weekly SMT. Prior to randomization, medical screening, standardized psychosocial questionnaires, mental stress testing, assessment of diet and physical activity, and exercise testing will be conducted. Additional biomarkers of risk will be assessed through measures of flow-mediated vasodilation, inflammation, platelet function, stress hormones, baroreflex, and heart rate variability.

Participants assigned to CR alone will engage in supervised exercise routines 3 times per week. Participants will be encouraged to maintain consistent exercise duration and effort throughout each session. Participants assigned to CR enhanced with SMT will engage in standard exercise-based cardiac rehabilitation and also receive weekly group SMT. At the conclusion of the 12-week intervention, participants will return for repeat assessments of stress and biomarker measures. At 6 months, 12 months, and annually up to 4 years participants will be contacted for information regarding major adverse cardiovascular events, other medical events and medication use.

Additionally a group of age, gender, and disease matched cardiac patients referred to CR, during the same time interval, but who elected not to participate in CR will form a non-randomized comparison group for cardiac events.

Overall, 164 participants were consented for study participation at Duke University Medical Center. Of these, 151 participants were randomized to either Standard Cardiac Rehabilitation or Enhanced Cardiac Rehabilitation. Post-intervention assessments were completed on 145 participants; 151 participants were available for intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Coronary Heart Disease (CHD)
* Eligibility for Cardiac Rehabilitation (CR) in North Carolina
* Capacity to give informed consent and follow study procedures

Exclusion Criteria:

* Received heart transplant
* LVEF < 30%
* Labile ECG changes prior to testing
* Currently using a pacemaker
* Resting BP > 200/120 mm Hg
* Left main disease > 50%
* Unable to comply with assessment procedures
* Unwilling or unable to be randomized to treatment groups
* Primary diagnosis of the following psychiatric disorders: schizophrenia, dementia, current delirium, or other psychotic disorder
* Current alcohol or substance abuse disorder
* Acute suicide risk
* Actively undergoing ongoing psychiatric treatment

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Blumenthal, PhD, Principal Investigator — Duke University; Alan Hinderliter, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina Hospitals - Meadowmont, Chapel Hill, North Carolina
  - Duke University Medical Center - Center for Living, Durham, North Carolina

REFERENCES:
- [Background] Blumenthal JA, Jiang W, Babyak MA, Krantz DS, Frid DJ, Coleman RE, Waugh R, Hanson M, Appelbaum M, O'Connor C, Morris JJ. Stress management and exercise training in cardiac patients with myocardial ischemia. Effects on prognosis and evaluation of mechanisms. Arch Intern Med. 1997 Oct 27;157(19):2213-23. PMID 9342998
- [Background] Rees K, Bennett P, West R, Davey SG, Ebrahim S. Psychological interventions for coronary heart disease. Cochrane Database Syst Rev. 2004;(2):CD002902. doi: 10.1002/14651858.CD002902.pub2. PMID 15106183
- [Background] Jones DA, West RR. Psychological rehabilitation after myocardial infarction: multicentre randomised controlled trial. BMJ. 1996 Dec 14;313(7071):1517-21. doi: 10.1136/bmj.313.7071.1517. PMID 8978226
- [Background] Frasure-Smith N, Lesperance F, Prince RH, Verrier P, Garber RA, Juneau M, Wolfson C, Bourassa MG. Randomised trial of home-based psychosocial nursing intervention for patients recovering from myocardial infarction. Lancet. 1997 Aug 16;350(9076):473-9. doi: 10.1016/S0140-6736(97)02142-9. PMID 9274583
- [Background] Balady GJ, Williams MA, Ades PA, Bittner V, Comoss P, Foody JM, Franklin B, Sanderson B, Southard D; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Epidemiology and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism; American Association of Cardiovascular and Pulmonary Rehabilitation. Core components of cardiac rehabilitation/secondary prevention programs: 2007 update: a scientific statement from the American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; the Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; and the American Association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2007 May 22;115(20):2675-82. doi: 10.1161/CIRCULATIONAHA.106.180945. Epub 2007 May 18. PMID 17513578
- [Background] Ades PA. Cardiac rehabilitation and secondary prevention of coronary heart disease. N Engl J Med. 2001 Sep 20;345(12):892-902. doi: 10.1056/NEJMra001529. No abstract available. PMID 11565523
- [Background] Wenger NK, Froelicher ES, Smith LK, Ades PA, Berra K, Blumenthal JA, Certo CM, Dattilo AM, Davis D, DeBusk RF, et al. Cardiac rehabilitation as secondary prevention. Agency for Health Care Policy and Research and National Heart, Lung, and Blood Institute. Clin Pract Guidel Quick Ref Guide Clin. 1995 Oct;(17):1-23. PMID 8595435
- [Background] Blumenthal JA, Babyak M, Wei J, O'Connor C, Waugh R, Eisenstein E, Mark D, Sherwood A, Woodley PS, Irwin RJ, Reed G. Usefulness of psychosocial treatment of mental stress-induced myocardial ischemia in men. Am J Cardiol. 2002 Jan 15;89(2):164-8. doi: 10.1016/s0002-9149(01)02194-4. PMID 11792336
- [Background] Blumenthal JA, Sherwood A, Babyak MA, Watkins LL, Waugh R, Georgiades A, Bacon SL, Hayano J, Coleman RE, Hinderliter A. Effects of exercise and stress management training on markers of cardiovascular risk in patients with ischemic heart disease: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1626-34. doi: 10.1001/jama.293.13.1626. PMID 15811982
- [Derived] Blumenthal JA, Sherwood A, Smith PJ, Watkins L, Mabe S, Kraus WE, Ingle K, Miller P, Hinderliter A. Enhancing Cardiac Rehabilitation With Stress Management Training: A Randomized, Clinical Efficacy Trial. Circulation. 2016 Apr 5;133(14):1341-50. doi: 10.1161/CIRCULATIONAHA.115.018926. Epub 2016 Mar 21. PMID 27045127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 164 participants were consented for study participation. Of these, 151 participants were randomized to either Standard Cardiac Rehabilitation or SMT-Enhanced Cardiac Rehabilitation. Post-intervention assessments were completed on 145 participants; 151 participants were available for intention-to-treat analysis.
Period: Overall Study
Arm/Group | SMT-Enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Started | 76 | 75
Completed | 73 | 72
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMT-enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.8) | 60.4 (10.6) | 61.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 45 | 51 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 23 | 40
  White | 58 | 51 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Composite Stress Score
Description: A global stress measure (mean rank), was the primary outcome combining the following components at baseline and following treatment: Beck Depression Inventory II, Spielberger Anxiety Inventory-State, General Health Questionnaire, PROMIS Anger Questionnaire, and Perceived Stress Scale. A range from 1 to 147 was present with higher scores suggestive of better function. The change in each individual scaled score is presented in primary outcome 2.
Time Frame: Baseline; 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Mean rank score
Arm/Group | SMT-enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
Mean rank score | 77.6 [71.5 to 83.7] | 67.5 [61.3 to 73.8]
Statistical Analysis 1: Comparison: SMT-enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; ANCOVA; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-18.7 to -1.5]

2. Primary Outcome: Change From Baseline to 12 Weeks in Individual Scaled Scores
Description: Beck Depression Inventory II: 21-item scale used to measure depression. Scores range from 0 to 63, with higher scores suggesting greater depressive symptoms.
  State-Trait Anxiety Inventory: 20-item scale which assess levels of state anxiety. Scores range from 20 to 80 with scores ≥40 suggesting clinically significant anxiety.
  General Health Questionnaire:12-item measure of general distress. Scores range from 0 to 36, with higher scores indicating greater emotional distress.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anger: 8-item scale which assesses anger. Scores range from 8 to 40, with higher scores indicating greater anger.
  Perceived Stress Scale: 10-item measure of general distress and perceived ability to cope. Scores range from 0 to 40, higher scores indicate greater stress.
Time Frame: Baseline; 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SMT-Enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
units on a scale
  Beck Depression Inventory-II | -3.5 [-5.0 to -2.1] | -2.6 [-4.1 to -1.2]
  Spielberger Anxiety Inventory-State | -5.6 [-7.4 to -3.7] | -2.6 [-4.5 to -0.7]
  General Health Questionnaire | -4.8 [-5.8 to -3.7] | -3.3 [-4.4 to -2.2]
  PROMIS Anger Questionnaire | -2.0 [-3.0 to -1.0] | -1.0 [-2.1 to 0.0]
  Perceived Stress Score | -4.2 [-5.4 to -3.0] | -2.6 [-3.9 to -1.3]
Statistical Analysis 1: Comparison: SMT-Enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; p < 0.05, ANCOVA

3. Secondary Outcome: Major Adverse Cardiovascular Events (MACE) - All Cause Death, MI, Cardiac Revascularization and Cardiovascular Hospitalization.
Description: Patients documented all medical encounters on an annual basis after enrollment. Medical records were reviewed, and events, categorized on the basis of American College of Cardiology/American Heart Association criteria. The following medical events were included: all-cause mortality, fatal and nonfatal myocardial infarction (MI), coronary or peripheral artery revascularization, stroke/transient ischemic attack, and unstable angina requiring hospitalization.
Time Frame: Baseline through Follow-up (median, 3.2 years)
Measure: Count of Participants; unit: Participants
Arm/Group | SMT-enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
Participants
  All cause mortality | 0 | 2
  MI | 1 | 6
  Stent/CABG | 9 | 11
  Stroke/TIA | 1 | 1
  Peripheral Revascularization | 1 | 3
  Angina Requiring Hospitalization | 2 | 2
Statistical Analysis 1: Comparison: SMT-enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; Log Rank; Cox Proportional Hazard = 0.47, 95% CI 2-sided [0.24 to 0.91]

4. Secondary Outcome: Change in High-sensitivity C-Reactive Protein
Description: High-sensitivity C-reactive protein was quantified by ELISA. Values >10 mg/L were truncated at 10 to account for acute inflammatory processes that may have skewed the distribution of this blood marker.
Time Frame: Baseline; 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Arm/Group | SMT-enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
mg/L | -0.9 [-1.4 to -0.5] | -0.4 [-0.9 to 0.0]
Statistical Analysis 1: Comparison: SMT-enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; p = .95, ANCOVA; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.14 to 1.17]

5. Secondary Outcome: Heart Rate Variability During Controlled Breathing (HRV-DB)
Description: Heart rate variability was obtained from beat-to-beat heart rate. Heart rate was assessed from R-R interval changes elicited during a 100-second controlled breathing task.
Time Frame: At 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: ms
Arm/Group | SMT-Enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
ms | 13.1 [-8.0 to 34.3] | 26.0 [5.5 to 46.5]
Statistical Analysis 1: Comparison: SMT-Enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; p = 0.99, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.22 to 0.46]

6. Secondary Outcome: Baroreflex Sensitivity
Description: Baroreflex sensitivity was obtained from beat-to-beat heart rate and blood pressure recorded from patients in the supine position with a Nexfin noninvasive blood pressure monitor.
Time Frame: At 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: ms/mm Hg
Arm/Group | SMT-Enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
ms/mm Hg | 0.47 [-0.39 to 1.33] | 0.93 [0.09 to 1.77]
Statistical Analysis 1: Comparison: SMT-Enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; p = 0.99, ANCOVA; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.78 to 1.74]

7. Secondary Outcome: Heart Rate Variability During Rest
Description: Heart rate variability was obtained from beat-to-beat heart rate. Heart rate was assessed from R-R interval changes elicited during 5 minutes of normal relaxed breathing
Time Frame: At 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: ln (ms^2)
Arm/Group | SMT-Enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Number analyzed (Participants) | 76 | 75
ln (ms^2)
  Low-frequency | 0.17 [-0.08 to 0.27] | 0.28 [0.04 to 0.51]
  High-frequency | 0.08 [-0.11 to 0.27] | 0.22 [0.03 to 0.41]
Statistical Analysis 1: Comparison: SMT-Enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; p = 0.99, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.22 to 0.46]
Statistical Analysis 2: Comparison: SMT-Enhanced Cardiac Rehabilitation vs Standard Cardiac Rehabilitation; Test type: Superiority; p = 0.99, ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.14 to 0.39]

ADVERSE EVENTS:
Arm/Group | SMT-enhanced Cardiac Rehabilitation | Standard Cardiac Rehabilitation
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

LIMITATIONS AND CAVEATS:
Comparison group was not randomized to non-CR; relatively small sample and few 'hard' end points over the follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No